CLINICAL TRIAL: NCT00569465
Title: Effects of Arginine and N-Acetylcysteine Administration on Nitric Oxide Production and Arterial Blood Pressure in Hypertensive Diabetic Patients.
Brief Title: N-Acetylcysteine and Arginine Administration in Diabetic Patients
Acronym: NACARGPAO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: End of the study
Sponsor: University of Turin, Italy (Other)
Responsible Party: Prof. Valentino Martina, University of Turin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EUDRACT 2004-004203-38
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2007-12-07 (Estimated); Status verified 2007-12

CONDITIONS: Type 2 Diabetes Mellitus; Hypertension
Keywords: nitric oxide; oxidative stress; diabetes; hypertension; endothelial dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Diabetes Mellitus | interventions — Arginine; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator)
  Interventions: Drug: Placebo
- B (Experimental)
  Interventions: Drug: Arginine; Drug: Acetylcysteine

INTERVENTIONS:
Drug: Arginine — 1200 mg, once a day
  Other Names: Zentrum
  Arms: B
Drug: Acetylcysteine — 600 mg twice a day
  Other Names: Acetilcisteina
  Arms: B
Drug: Placebo — 3 vials a day
  Arms: A

SUMMARY:
It has been demonstrated that the nitric oxide production is reduced in type 2 diabetic patients and that cardiovascular complications represent 80% of the causes of death in these patients. As nitric oxide is able to reduce platelet aggregation, increase the relaxation of smooth muscle cells, and reduce plasminogen activator inhibitor-1 and endothelin, we hypothesized that nitric oxide deficiency is responsable for the cardiovascular disease in type 2 diabetes mellitus. Arginine and N-acetylcysteine, precursor and enhancer of the nitric oxide synthesis respectively, are able to increase nitric oxide production.

Aim of the study is to evaluate the effect of arginine and N-acetylcysteine administration on arterial blood pressure and different metabolic parameters in patients with type 2 diabetes mellitus and hypertension.

Subjects and methods. 24 male subjects, randomly divided in two groups, will be studied. These subjects will undergo a treatment with arginine (1200 mg once a day) plus N-acetylcysteine (600 mg twice a day) or placebo for six months. Basal and final evaluations include:

* general examination
* ABPM (ambulatory blood pressure monitoring)
* HbA1c, total-cholesterol, HDL-cholesterol, LDL-cholesterol, oxidized LDLs, triglycerides, reduced/oxidized glutathione ratio in red blood cells, nitrites/nitrates, asymmetrical and symmetrical dimethyl-arginine, nitrotyrosine, arginine, homocysteine, C-reactive protein, interleukin-6, tumor necrosis factor-α, intercellular and vascular-cell adhesion molecules, plasminogen activator inhibitor-1 and fibrinogen
* the ultrasound assessment of the intima-media thickness after endothelium-dependent flow-mediated vasodilation of the brachial artery

Expected results. Increase of nitric oxide production and reduction of arterial blood pressure and oxidative parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects
* Age between 40 and 70 years
* Type 2 diabetes mellitus and hypertension
* Mean 24h arterial blood pressure after the wash-out period: systolic >136mmHg and/or diastolic >86 mmHh
* Written informed consent

Exclusion Criteria:

* Female subjects
* Mean 24h arterial blood pressure after the wash-out period: systolic >180 mmHg and/or diastolic >110 mmHg
* Secondary hypertension
* Significative cardiovascular complications of diabetes
* Cancer or severe systemic, hepatic, pulmonary, cardiovascular or diseases
* Actual treatment with nitrates, acetylcysteine or arginine
* Acetylcysteine hypersensitivity
* Psychiatric disturbs, abuse of drugs or alcohol
* Low compliance
* Absence of written informed consent

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-01; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
arterial blood pressure decrease | 6 months

SECONDARY OUTCOMES:
oxidative parameters decrease | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Valentino Martina, MD, Principal Investigator — University of Turin, Italy
Locations (1):
- "San Giovanni Battista" Hospital of Turin, Turin, Turin, Italy